CLINICAL TRIAL: NCT07203820
Title: The Effect of Ready-made Picture Template Coloring Activity on Children's Anxiety and Fear Before Circumcision: A Randomized Controlled Trial
Brief Title: Children's Anxiety and Fear Before Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Maksude YILDIRIM, Assistant Professor, Adiyaman University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HRÜ/24.21.05
Record Dates: First submitted 2025-01-15; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Fear
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ready-Made Picture Template Painting Activity (Experimental): The child will be asked to go to the child with the ready-made picture template and coloring pencils and color the given picture with the colors they want.
  Interventions: Behavioral: Ready-Made Picture Template Painting Activity
- Control group (No Intervention): No procedures other than routine procedures performed in the hospital will be applied to the children in this group

INTERVENTIONS:
Behavioral: Ready-Made Picture Template Painting Activity — The purpose of the study will be explained to the children and their parents before the painting process and verbal and written consent will be obtained from the parents who agree to participate in the study. The child will be asked to go to the child with the ready-made picture template and coloring pencils and color the given picture with the colors they want. Children's anxiety will be assessed using the Children's State Anxiety (CSA) and their fears will be assessed using the Children's Fear Scale (CFS) based on both mother's and child's reports before painting and after the painting process is completed (half an hour after the first measurement).
  Arms: Ready-Made Picture Template Painting Activity

SUMMARY:
This study was planned as a randomized controlled trial to investigate the effect of ready-made picture template coloring activity on children's anxiety and fear before circumcision. Data is planned to be collected between November 2024 and February 2025 with children between the ages of 5-10 who are planned to be circumcised in a hospital in the Southeastern Anatolia Region. The study consists of painting and control groups. The group in which the participants will be included will be determined by the stratified randomization method. The anxiety status of the children in the painting and control groups will be evaluated using the Children's State Anxiety (CSA) and their fears will be evaluated using the Children's Fear Scale (CFS) based on the reports of both the mother and the child before and after painting. Data collection will be completed before the child is circumcised.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 5-10,
* who are planned to be circumcised,
* who are not in pain, and
* whose parents approve of participating in the study will be included in the study.

Exclusion Criteria:

* Children with mental retardation,
* bleeding disorders, and
* traumatic experiences such as death and divorce in the last year will not be included in the study.

Ages: 5 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Boys circumcised in Turkey
Enrollment: 50 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Children's State Anxiety | 4 months
  The scale aims to measure the situational anxiety of children in the 4-10 age group
Children's Fear Scale | 4 months
  The scale, which evaluates children's odors with photographs containing facial muscle changes, can be used by children, families, or researchers

CONTACTS AND LOCATIONS:
Locations (1):
- Harran University, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No